CLINICAL TRIAL: NCT00198887
Title: Operations Research to Improve Newborn Health and Survival in the (INHP-II) Area of CARE/India
Brief Title: Operations Research to Improve Newborn Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: H.22.02.08.30.A2
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Pregnancy Complications
Keywords: newborn; operations research; newborn survival; Neonatal illness/mortality; Delivery complications
MeSH Terms: conditions — Pregnancy Complications

INTERVENTIONS:
Procedure: Operations research

SUMMARY:
This study is designed to look at how operations are carried out in relation to improving the health and survival of newborn babies in India.

DETAILED DESCRIPTION:
The proposed study aims to evaluate the impact of a basic package of obstetric and neonatal care practices implemented by CARE-India as part of their ten-year, two-phase Integrated Nutrition and Health Program (INHP). Building on the lessons learned from the Integrated Nutrition and Health Project I (INHP I) in seven Indian states during 1996-2001, CARE-India has designed INHP II, which focuses on six technical interventions. CARE-India aims to implement this program in 100,000 villages across eight states of India by the year 2006. One of the technical interventions is a focused package of newborn care to be implemented at the community level to improve the health and survival of the newborns, including improvements in care-seeking for maternal and newborn conditions. The services and behaviors promoted include:

1. antenatal care,
2. iron-folate supplementation,
3. tetanus toxoid vaccination,
4. maternal nutrition and rest,
5. birth planning,
6. essential newborn care,
7. immediate and exclusive breastfeeding,
8. prevention of hypothermia,
9. aseptic cord care, and
10. identification and referral of cases with danger signs for both pregnancy/delivery complications and newborn conditions.

The services are provided by first-line community-based health workers.

CARE-India invited Johns Hopkins Bloomberg School of Public Health (JHBSPH) to help evaluate their newborn program in an operations research mode. JHBSPH's role is limited to assisting CARE with the design and evaluation of newborn intervention.

ELIGIBILITY:
Inclusion Criteria:

* Newborn

Exclusion Criteria:

* Infant/child

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59651 (Actual)
Dates: Start 2003-01; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Neonatal mortality rate

SECONDARY OUTCOMES:
Cost of delivering the intervention, per newborn
Changes in behavioral indicators
Change in program coverage

CONTACTS AND LOCATIONS:
Overall Officials: Mathuram Santosham, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- King George's Medical College, Lucknow, Uttar Pradesh, India